CLINICAL TRIAL: NCT07405645
Title: Stereotactic MRI-guided Focused Ultrasound Mesencephalotomy for Pain Palliation in Head, Neck, & Brachial Cancer
Brief Title: Stereotactic MRI-guided Focused Ultrasound Mesencephalotomy
Acronym: MRg-FUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Focused Ultrasound Foundation (Other)
Responsible Party: Principal Investigator, Jeff Elias, MD, Professor of Neurological Surgery, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSR180040-1
Record Dates: First submitted 2026-01-22; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Head Neck Cancer; Squamous Cell Cancer of Head and Neck (SCCHN); Cancer Pain
Keywords: cancer pain; mesencephalotomy; focused ultrasound
MeSH Terms: conditions — Head and Neck Neoplasms; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Group Assignment (Experimental): Single Group Assignment
  Interventions: Device: ExAblate Neuro

INTERVENTIONS:
Device: ExAblate Neuro — Exablate Neuro uses focused ultrasound waves to precisely target and ablate tissue deep within the brain with no incisions or implants. The treatment is done under Magnetic Resonance Imaging (MRI) guidance for real time treatment monitoring.

SUMMARY:
This phase 1 multi-site study investigates the safety and initial effectiveness of focused ultrasound lesioning of the contralateral mesencephalon for severe, opioid-resistant pain associated with head and neck cancer and brachial cancer.

DETAILED DESCRIPTION:
This phase 1 study investigates the safety and initial effectiveness of focused ultrasound lesioning of the contralateral mesencephalon for severe, opioid-resistant pain associated with head, neck, and brachial cancer.

Safety: To evaluate the incidence and severity of adverse events associated with unilateral stereotactic focused ultrasound mesencephalotomy.

Efficacy: To determine the level or degree of pain relief in the head, neck, and brachial regions using validated numeric pain scales and patient-reported measures of pain.

The rationale for this proposed Phase 1 study is based upon:

1. The pain associated with head, neck, and brachial cancer is one of the most severe and difficult conditions because it is:

   * notoriously refractory to medical therapies,
   * localized to the highest regions of the neural axis and is thus not amenable to traditional surgical options like intrathecal opioids or spinal cordotomy, and
   * affects them during the terminal stages of life.
2. Stereotactic mesencephalotomy, targeted to the confluence of the spinoreticular and spinothalamic tracts, has been associated with pain relief from malignancy, but historical stereotactic methods lacked precision to reduce morbidity for routine adoption.
3. Focused ultrasound has been demonstrated to be a precise stereotactic lesioning modality, and the technique can be performed without incisions or craniotomy. Continuous closed-loop monitoring of the thermal ablation process with MRI has yielded lesion accuracies consistently < 1 millimeter.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, between 18 and 85 years, inclusive
2. Subjects with head, neck, or brachial cancer, including one of the following:

   * Cancer that arises in the head and neck region: nasal cavity, sinuses, lips, mouth, salivary glands, throat, or larynx (typically squamous cell carcinoma)
   * Cancer occurring in the nasopharynx, skin, thyroid gland, and eye
   * Cancer involving the brachial region including brachial plexus, upper lung apex, and Pancoast tumors.
   * Lymphoma
   * Sarcoma
3. Craniofacial, cervical, or brachial pain related to the cancer that meets all of the following criteria:

   * Severe defined by: Worst NPRS score of ≥ 5 out of 10 at current visit and the subject reports having a similar level of pain for at least the past two months.
   * Pain is medication-refractory to all three tiers of the WHO cancer pain ladder. Thus, adequate trials of at least 3 prescription medications that will include a 'weak' and a 'strong' opioid. An adequate medication trial is defined as a therapeutic dose of each medication without sufficient effect.
   * Duration of greater than 3 months.
4. Mesencephalon contralateral to the pain can be targeted by the ExAblate Neuro device. The region of the mesencephalon must be apparent on MRI. Additional MRI sequences including inversion-recovery and DTI may be utilized to refine the target.
5. Subjects who are able and willing to give consent and able to attend all study visits
6. Subjects who are able to communicate sensations during the focused ultrasound treatment

Exclusion Criteria:

1. Idiopathic trigeminal neuralgia
2. Trigeminal neuropathic pain from trauma, infection, or iatrogenic
3. Post-herpetic neuralgia
4. Headache syndromes like migraine, cluster headache
5. Temporomandibular joint syndrome
6. Atypical facial pain or pain related to a somatoform disorder
7. Subjects deemed poor candidates by a multidisciplinary team of cancer and palliative care clinicians:

   1. Subject deemed by their oncologist to have limited life expectancy for outcome assessment. At least 3 months life expectancy is required to obtain the primary efficacy outcome measure.
   2. Significant clinician concern about reliability of subject-reported information, such as subject in active process of seeking disability for neuropathic pain
   3. Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-V as manifested by one (or more) of the following occurring within a 12 month period: Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (such as repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; or neglect of children or household). Recurrent substance use in situations in which it is physically hazardous (such as driving an automobile or operating a machine when impaired by substance use)
   4. Recurrent substance-related legal problems (such as arrests for substance related disorderly conduct)
   5. Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (for example, arguments with spouse about consequences of intoxication and physical fights).
8. Subjects with active psychiatric illness will be excluded. For the purpose of this study, active psychiatric illness includes:

   1. Exhibiting current suicide ideation and/or a history of suicide attempt within past 2 years
   2. been hospitalized for the treatment of a psychiatric illness within the past 2 years
   3. received transcranial magnetic stimulation for depression treatment
   4. received electroconvulsive therapy for depression
   5. any presence or history of psychosis
9. Subjects with unstable cardiac status including:

   1. Unstable angina pectoris on medication
   2. Subjects with documented myocardial infarction within six months of protocol entry
   3. Significant congestive heart failure defined with ejection fraction < 40
   4. Subjects with unstable ventricular arrhythmias
   5. Subjects with atrial arrhythmias that are not rate-controlled
10. Severe hypertension (diastolic BP > 100 on medication)
11. Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
12. On medications that increases the bleeding risk, based on the published guidelines which are currently recognized by the American Society of Regional Anesthesia and Pain Medicine, American Academy of Pain Medicine and the North American Neuromodulation Society (Reg Anesth Pain Med 2015;40: 182-212); specifically:

    1. Aspirin or another antiplatelet medication (clopidogrel, prasugrel, ticlopidine, abiciximab) for the last 7 days prior to treatment.
    2. Oral, subcutaneous or intravenous anticoagulant medications, such as oral vitamin K inhibitors for the last 7 days, non-vitamin K inhibitor oral anticoagulant (dabigatran, apixaban, rivaroxaban) for the last 72 hours.
    3. Intravenous or subcutaneous heparin-derived compounds for the last 48 hours.
13. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hours of total table time.)
14. Subjects participating or have participated in another pain management clinical trial in the last 30 days
15. Subjects with risk factors for intraoperative or postoperative bleeding from a documented coagulopathy or if their serum coagulation studies (platelet count, PT, PTT, and INR) exceed the institutional laboratory limits.
16. Subjects with brain tumors or any significant intracranial mass that impedes the acoustic beam. Subjects with cerebral metastasis may be included if the lesion(s) do not affect the FUS treatment.
17. Any illness that in the investigator's opinion preclude participation in this study
18. Pregnancy or lactation
19. Legal incapacity or limited legal capacity
20. Subjects with a deep brain stimulation implant
21. Skull density ratio, calculated from the baseline noncontrasted head CT, is less than 0.4
22. History of hemorrhagic stroke or cerebrovascular event within the past year of treatment exhibiting incomplete resolution
23. Subjects whose primary pain is other than craniofacial or brachial neuropathic pain.
24. Patients deemed high risk because of their airway for the procedure as evaluated by anesthesia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Outcome | Intervention through 6 months
  Safety as assessed from adverse event reporting.
Primary Efficacy Outcome | 24 hours before (baseline) and at 3 months following unilateral FUS mesencephalotomy
  To compare the change of WORST pain experienced. 11-point Numeric Pain Rating Scale (NPRS)

SECONDARY OUTCOMES:
Secondary Outcomes | baseline to 3 months post-treatment
  Patient Global Impression of Change and the Pain Domain from the PROMIS Inventory including items for intensity, quality, behavior and interference.

CONTACTS AND LOCATIONS:
Overall Officials: William J Elias, MD, Principal Investigator — University of Virginia
Locations (6):
- United States (6):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Weill Cornell Medicine, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No